CLINICAL TRIAL: NCT05668026
Title: Administration of the BCL-2 Antagonist, Venetoclax, to Promote Apoptosis of HIV-infected Cells and Reduce the Size of the HIV Reservoir: An Investigator-initiated Phase I/IIb Clinical Trial in People Living With HIV on Antiretroviral Therapy
Brief Title: Administration of Venetoclax to Promote Apoptosis of HIV-infected Cells and Reduce the Size of the HIV Reservoir Among People Living With HIV on ART
Acronym: AMBER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: The Peter Doherty Institute for Infection and Immunity (Other); Walter and Eliza Hall Institute of Medical Research (Other); The Alfred (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMB-001; 2022-001677-31 (EudraCT Number)
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-04

CONDITIONS: HIV-1-infection
Keywords: HIV-1; bcl-2 inhibitor; venetoclax; anti-apoptotic protein
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: Dose-escalation study and an expansion cohort based on dose-limiting toxicities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Experimental): Study participants will receive venetoclax daily for 14 days followed by 21 days off defined as one cycle. This dosing will then be repeated for two additional cycles.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — In this study participants will receive venetoclax 200 mg, 400 mg or 800 mg once daily for 14 days in the dose-escalation phase. In the expansion cohort, the selected max-tolerated dose will be given for three cycles, each consisting of venetoclax daily for 14 days followed by 14 days off.

SUMMARY:
In summary, there is a compelling rationale for investigating venetoclax as an intervention to sensitise virus-expressing cells to apoptosis and thereby reduce the size of the latent HIV reservoir. While this concept may ultimately need to be tested in the setting of concomitant latency reversal, the investigators propose to initially establish the safety of venetoclax in PLWH on ART. The investigators will use this study to also investigate effects of venetoclax monotherapy on proapoptotic pathways, immune effector function and HIV persistence in PLWH on ART and through these studies establish the rationale for subsequent studies testing venetoclax in combination with an LRA.

DETAILED DESCRIPTION:
Despite the great success of antiretroviral therapy (ART) in suppressing HIV replication, treatment for people living with HIV (PLWH) is lifelong and there is no cure. The main reason ART is unable to cure HIV is the persistence of HIV in a latent form in long-lived and proliferating CD4+ T-cells [1]. One strategy to eliminate latently infected cells, referred to as shock and kill, is by activating HIV expression in latently cells with the aim of eliminating infected cells through either virus-induced apoptosis or immune-mediated killing. This has been tested in several clinical trials using various latency-reversing agents (LRAs), but although these studies provided evidence that HIV latency can be disrupted in PLWH on ART, this did not lead to a reduction in the frequency of latently infected cells.

Multiple studies have now demonstrated that not all infected cells that persist on ART have truly latent virus. In other words, residual low level transcription can persist on ART, measured as persistent detection of either cell associated HIV RNA or expression of p24 protein. These transcriptionally or translationally active cells are often more commonly found in tissue than in blood and is now referred to as the ''active reservoir''. For these cells, it is possible that expression of viral proteins could potentially either protect from or enhance cell death. It remains unclear why or how these cells can persist on ART, given their expression of viral proteins.

A key barrier to effective elimination of infected cells, either the latent or active reservoir, may be a reduced susceptibility to killing of infected cells that persist on ART. Previous studies highlighted the considerable heterogeneity among subsets of CD4+ T cells in susceptibility to apoptosis [8, 9] and one study also showed that increased sensitivity to killing of infected cells may play a role in the exceptional control of HIV without ART seen in elite controllers [10]. By performing RNA sequencing of latently infected CD4+ T cells that survived co-culture with HIV-specific cytotoxic T cells (CTLs), Ren et al recently demonstrated that over-expression of the pro-survival factor B cell lymphoma 2 (BCL-2) is a prominent feature of cells that are resistant to killing and that the inducible HIV reservoir was disproportionately present in BCL-2hi CD4+ T cells.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Age 18-65 years, both included
* Receiving combination ART for at least 2 years and being on the same ART regimen for at least 4 weeks at the screening visit
* HIV-1 plasma RNA <50 copies/mL for >2 years (documented on at least 2 occasions within the 2 years) and <20 copies/mL at screening. Episodes of a single HIV plasma RNA 50-500 copies/mL will not exclude participation if the subsequent HIV plasma RNA was <50 copies/mL
* CD4+ T cell count >500 cells/yL at screening and at least two CD4+ T cell counts >500 cells/yL in the 24 months prior to screening
* Ability and willingness to provide informed consent and to continue ART throughout the study
* For potential study participants who anticipate receiving a SARS-CoV-2 vaccine within the study period, enrolment and commencement of study therapy will be postponed until 4 weeks after completing SARS-CoV-2 vaccination, whereas screening procedures can be initiated before or concurrently with SARS-CoV-2 vaccination.
* A female, may be eligible to enter and participate in the study if she:

  * Is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
  * Is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:

    * Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all study medications
    * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year
    * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject
    * Approved hormonal contraception (Where other medications to be used in the study (e.g., efavirenz and darunavir) are known, or are likely, to significantly interact with systemic contraceptives, resulting in decreased efficacy of the contraceptive, then alternative methods of non-hormonal contraception are recommended)
    * Any other method with published data showing that the expected failure rate is <1% per year
    * Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of study therapy.
* All participants must agree not to participate in a conception process (e.g. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization, egg donation) during the study
* Heterosexually active male if they are

  * willing to use an effective method of contraception (anatomical sterility in self that is confirmed prior to study entry) or
  * agree on the use of an effective method of contraception with an effective failure rate of < 1% by his partner (hormonal contraception, intra-uterine device (IUD), or anatomical sterility) from the day prior to the first dose and for at least 2 weeks after discontinuation of study drug.

Exclusion Criteria:

* Current or previous use of a BCL-2 antagonist or other pro-apoptotic agent used as cancer therapy
* Any concomitant disease where venetoclax treatment is indicated
* Current use of any moderate or strong CYP3A4 inhibitors (such as ketoconazole, voriconazole, posaconazole, itraconazole, ritonavir, cobicistat and clarithromycin)
* Current use of any HIV protease inhibitor (due to CYP3A4 inhibition)
* Current use of any strong inhibitor of the P-gp drug efflux pump (this includes cobicistat, ritonavir, azithromycin and clarithromycin)

  * current use of drugs that are P-gp substrates (such as TDF, TAF and dolutegravir) is allowed but will require venetoclax dosing at least 6 hours after intake of those drugs
  * for study participants receiving TDF or TAF we will perform enhanced renal monitoring by quantifying estimated glomerular filtration rate (eGFR) at each study visit during venetoclax administration
* Current use of strong CYP3A4 inducers (such as carbamazepine, phenytoin, rifampicin and St. John's wort); moderate CYP3A4 inducers (such as bosentan, efavirenz, etravirine, modafinil and nafcillin) may be used but should be avoided as much as possible
* Receipt of immunomodulating agents (excluding immunisation) or systemic chemotherapeutic agents within 28 days prior to study entry
* Any other current or prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study
* Known hypersensitivity to the components of venetoclax or its analogues
* Any significant acute medical illness in the past 4 weeks
* Any evidence of an active AIDS-defining opportunistic infection
* Individuals who intend to modify their ART regimen within the study period
* Current or recent gastrointestinal disease or gastrointestinal surgery that may impact the absorption of the investigational drug
* Active alcohol or substance use that, in the Investigator's opinion, will prevent adequate compliance with study therapy or procedures
* Unable or unwilling to adhere to protocol procedures
* History of malignancy or transplantation, excluding adequately treated basal cell carcinoma
* Co-infection with hepatitis B or C (Individuals with prior hepatitis C infection that is now cleared are eligible for enrolment)
* Impaired liver function with AST or ALT >3 times upper limit of normal
* Severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Impaired renal function with estimated creatinine clearance (eGFR) <50 mL/min
* Significant cardiac dysfunction
* Women who are pregnant or breastfeeding or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy as specified in the inclusion criteria
* The following laboratory values at screening (lab tests may be repeated, as clinically indicated, to obtain acceptable values before failure at screening is concluded but supportive therapies are not to be administered within the week prior to screening tests)

  * Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN)
  * eGFR <50 mL/min
  * Platelet count ≤100 x109/L
  * Absolute neutrophil count ≤1.5x109/L
  * Haemoglobin <10,0 g/dL
  * Total lymphocyte count <800 cells/yL
  * CD4+ T cell count <500 cells/yL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of venetoclax in PLWH on ART | 0-140 days
  Incidence of treatment-emerging adverse events (AEs) >=grade 3 probably or definitely related to study treatment.
  Safety defined as all other treatment-emerging AEs, graded according to severity and assessed as either not related or possibly, probably or definitely related to study treatment.

SECONDARY OUTCOMES:
To determine the effect of venetoclax on HIV persistence in PLWH on ART | 0-140 days
  The size of the HIV-1 reservoir using the Intact Proviral DNA Assay (IPDA)
To determine the effect of venetoclax on proapoptotic pathways in PLWH on ART | 0-140 days
  Activation of pro-apoptotic pathways using cytometry by time of flight (CyTOF) and/or single cell RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Rasmussen, Principal Investigator — Department of Infectious Diseases, Aarhus University Hospital; Sharon R Lewin, Principal Investigator — The Peter Doherty Institute for Infection and Immunity (Doherty Institute), University of Melbourne
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark